CLINICAL TRIAL: NCT01941992
Title: Role of SAMITAL® in Prevention and Treatment of Oral Mucositis in Patients Treated With Chemo-radiation (CT/RT)for Head-and-neck Squamous Cell Carcinomas. A Double-blind, Phase 2 Placebo Controlled, Randomized Trial.
Brief Title: Role of SAMITAL® in the Relief of Chemo-radiation (CT-RT) Induced Oral Mucositis in Head and Neck Cancer Patients
Acronym: ROSAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IOV-HN-1-2012 ROSAM; 2012-002046-20 (EudraCT Number)
Record Dates: First submitted 2013-08-08; First posted 2013-09-13 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Head-and-neck Squamous Cell Carcinoma; Oral Mucositis
Keywords: head and neck; Squamous Cell Carcinoma; oral mucositis; Chemo-radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis; Carcinoma, Squamous Cell | interventions — samital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SAMITAL® sachets, oral suspension (Experimental): SAMITAL® sachets for oral suspension, 20 mL, four times a day.
  Interventions: Drug: SAMITAL®
- Placebo sachets (Placebo Comparator): Placebo sachets for oral suspension, 20 mL, four times a day.
  Interventions: Drug: Placebo sachets

INTERVENTIONS:
Drug: SAMITAL®
  Arms: SAMITAL® sachets, oral suspension
Drug: Placebo sachets
  Arms: Placebo sachets

SUMMARY:
The purpose of this study is to:

* evaluate the activity of SAMITAL in reducing the incidence of severe mucositis in head-and-neck cancer patients undergoing chemo-radiotherapy.
* assess tolerability of SAMITAL and the impact on patients reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinomas of the head-and-neck
* Eligible primary tumor sites: oral cavity, oropharynx, larynx, hypopharynx
* Stage III or IV disease without evidence of distant metastases
* Patients candidate to definitive concurrent chemo-radiotherapy or induction chemotherapy followed by chemo-radiotherapy
* Age ≥ 18 years
* Karnofsky Performance Status ≥70
* Life expectancy ≥6 months
* Able to swallow and retain oral medication
* Good state of dentition
* Patients must be available for treatment and follow-up
* Confirmation of adequate contraception use by the patient and/or partner
* Signed informed consent

Exclusion Criteria:

* Previous radiotherapy of the oral cavity, and/or oropharynx, larynx, hypopharynx
* Serious co-morbidities: uncontrolled heart disease, heart failure within 6 months prior to study participation, history of serious neurological and/or psychiatric abnormalities.
* Chronic administration of steroids or immunosuppressants
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with Grade III or IV of mucositis assessed by the WHO mucositis scale, developing at any time during the whole study period. | Within 19 weeks after starting Radiotherapy

SECONDARY OUTCOMES:
Incidence of adverse events assessed by NCI-Common Terminology Criteria for Adverse Effects (CTCAE version 4.0) | Within 19 weeks after starting Radiotherapy

OTHER OUTCOMES:
Quality of life assessed by European Organization for Research and Treatment of Cancer quality of life core questionnaire (EORTC QLQ-C30) and specific head and neck module (QLQ-H&N35) | Within 19 weeks after starting Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Loreggian, MD, Principal Investigator — Radiotherapy Department, Istituto Oncologico Veneto
Locations (1):
- Radiotherapy Department, Istituto Oncologico Veneto, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fasanaro E, Del Bianco P, Groff E, Riva A, Petrangolini G, Busato F, Stritoni P, Scarzello G, Loreggian L, De Salvo GL. Role of SAMITAL in the Prevention and Treatment of Chemo-Radiotherapy-Induced Oral Mucositis in Head and Neck Carcinoma: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Trial (ROSAM). Cancers (Basel). 2022 Dec 15;14(24):6192. doi: 10.3390/cancers14246192. PMID 36551677